CLINICAL TRIAL: NCT05627999
Title: Trans-anal Eco-doppler Evaluation of Haemorrhoidal Vascularization After Percutaneous Hemorrhoidal Artery Embolization. A Pilot Study.
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Ospedale Civile Ca' Foncello (Other)
Responsible Party: Principal Investigator, Giulio Aniello Santoro, Surgeon, Ospedale Civile Ca' Foncello
Other Study IDs: OCCaFoncello
Record Dates: First submitted 2022-11-16; First posted 2022-11-28 (Actual); Last update posted 2023-02-27 (Actual); Status verified 2023-02

CONDITIONS: Haemorrhoidal Bleeding

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- patients candidate to the haemorrhoidal artery embolization: Consecutive patients assessed at the Division of General Surgery 1, Treviso Regional Hospital, from October to December 2021 and candidate to the haemorrhoidal artery embolization were included in the study. Indications to the procedure were symptomatic hemorrhoidal disease (French bleeding score [FBS] > 4), Goligher's classification score II or III, age >18 years, failure of non-operative management (change life style, dietary modification, supplemental fibers for constipation, over-the-counter treatments). Signed informed and research consents were obtained. Exclusion criteria were age < 18 years, Goligher prolapse score IV, pregnancy, previous haemorrhoidal surgery, inflammatory bowel disease. Use of anticoagulant or antiaggregant was not considered an exclusion criteria [stecca].
  Interventions: Procedure: doppler endoanal ultrasound

INTERVENTIONS:
Procedure: doppler endoanal ultrasound — The primary aim was to assess the reduction in the blood supply by comparing the hemorrhoidal arterial systolic peak (overall and sectorial) before and after Emborrhoid.

SUMMARY:
To evaluate the usefulness of endoanal ultrasound in the evaluation of emorrhoidal artery embolization outcomes

DETAILED DESCRIPTION:
Haemorrhoidal artery embolization (Emborrhoid) is a novel method for the treatment of haemorrhoids. Through the catheterization of the femoral artery and a selective angiogram of the inferior mesenteric artery, embolic agents are delivered to occlude the SRA. Despite the technical success rate has been reported to reach 93%-100%, clinical success ranges between 63% and 94% with rebleeding occurring in 13.6% of cases due to the presence of a significant MRA in 24% of cases [BIBLIO} . There is no data in the literature on how the arterial flow changes after the treatment.

The primary aim of the present study was to assess the reduction in the blood supply by comparing the hemorrhoidal arterial systolic peak before and after Hemborrhoid by using endoanal ultrasound (EAUS) combined with doppler. The secondary aim was to evaluate if a relation exists between the reduction and the efficacy of this treatment by the Hemorrhoidal Bleeding Score.

ELIGIBILITY:
Inclusion Criteria:

* symptomatic hemorrhoidal disease (French bleeding score [FBS] > 4), Goligher's classification score II or III, age >18 years, failure of non-operative management (change life style, dietary modification, supplemental fibers for constipation, over-the-counter treatments).

Exclusion Criteria:

* age < 18 years, Goligher prolapse score IV, pregnancy, previous haemorrhoidal surgery, inflammatory bowel disease.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Consecutive patients assessed at the Division of General Surgery 1, Treviso Regional Hospital, from October to December 2021 and candidate to the haemorrhoidal artery embolization were included in the study.
Sampling Method: Non-Probability Sample
Enrollment: 10 (Estimated)
Dates: Start 2023-01-19 (Actual); Primary Completion 2023-02-19 (Actual); Study Completion 2023-03-20 (Estimated)

PRIMARY OUTCOMES:
the reduction in the blood supply | one month
  The primary aim was to assess the reduction in the blood supply by comparing the hemorrhoidal arterial systolic peak (overall and sectorial) before and after Emborrhoid.

SECONDARY OUTCOMES:
correlate the systolic peak reduction at the doppler analysis with the patients' symptoms improvement. | one month

CONTACTS AND LOCATIONS:
Locations (1):
- Ospedale Ca Foncello, Treviso, Italy

IPD SHARING:
Plan to Share IPD: Yes
A prospective observational pilot study was conducted. The primary aim was to assess the reduction in the blood supply by comparing the hemorrhoidal arterial systolic peak (overall and sectorial) before and after Emborrhoid. The secondary aim was to evaluate the efficacy of this treatment by the Hemorrhoidal Bleeding Score and to correlate the systolic peak reduction at the doppler analysis with the patients' symptoms improvement.
Supporting Information: Study Protocol, SAP